CLINICAL TRIAL: NCT06162468
Title: Single-arm Intervention Trial of the Feasibility of Endoscopic Ultrasound-guided Pancreatic Cyst Chemoablation (EUS-PCA) Using Gemcitabine and Paclitaxel for Intraductal Papillary Mucinous Neoplasms (IPMN) in Two New Zealand Tertiary Interventional Endoscopy Centres
Brief Title: Feasibility Trial of EUS-PCA in IPMN Pancreatic Cysts
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Auckland, New Zealand (Other)
Collaborators: Gut Cancer Foundation, New Zealand (Unknown); North Shore Hospital, New Zealand (Other); Waikato Hospital (Other)
Responsible Party: Principal Investigator, Michael Jameson, Associate Professor, University of Auckland, New Zealand
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTNZ-2022-06
Record Dates: First submitted 2023-11-20; First posted 2023-12-08 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Intraductal Papillary Mucinous Neoplasm of Pancreas
MeSH Terms: conditions — Pancreatic Intraductal Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Intervention Model Description: A single-arm trial of the feasibility of endoscopic ultrasound-guided pancreatic cyst chemoablation (EUS-PCA) using gemcitabine and paclitaxel for intraductal papillary mucinous neoplasms (IPMN) in two New Zealand tertiary interventional endoscopy centres.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-arm (Experimental): Gemcitabine 19 mg per 1 ml of estimated cyst fluid + paclitaxel 3 mg per 1 ml of estimated cyst fluid + 0.9% sodium chloride solution, given as a single administration
  Interventions: Procedure: Endoscopic ultrasound-guided pancreatic cyst chemoablation (EUS-PCA) using gemcitabine and paclitaxel

INTERVENTIONS:
Procedure: Endoscopic ultrasound-guided pancreatic cyst chemoablation (EUS-PCA) using gemcitabine and paclitaxel — EUS-PCA using gemcitabine and paclitaxel

SUMMARY:
The goal of this single-arm intervention trial is to determine the feasibility of implementing endoscopic ultrasound-guided pancreatic cyst chemoablation (EUS-PCA) using gemcitabine and paclitaxel for intraductal papillary mucinous neoplasms (IPMN) in two New Zealand tertiary interventional endoscopy centres.

DETAILED DESCRIPTION:
Early detection and treatment of pancreatic premalignant lesions, most commonly IPMN, may be the best current strategy to prevent invasive pancreatic cancer. The rates of IPMN progression to invasive cancer range from 7 to 25% at 10 years, depending on risk characteristics. The feasibility and safety of EUS-PCA has been demonstrated in studies, including smaller randomised trials, totaling about 140 participants. EUS-PCA with the chemotherapy drugs being used in this trial has been implemented in several major international centres due to its potential for the minimally-invasive prevention of invasive pancreatic cancer, though it has never been compared to surgery in a clinical trial.

This single-arm intervention trial will evaluate the feasibility of implementing endoscopic ultrasound-guided pancreatic cyst ablation (EUS-PCA) for IPMN in interventional endoscopy units in two New Zealand tertiary centres. Doing so in a clinical trial is consistent with the recommendation of an international expert panel to implement EUS-PCA in the context of a research trial.

A previous US trial reported a complete response rate at 12 months of 59%, with response maintained or further improved at 3 years. Of those with complete response, >95% of patients had not relapsed a median of 6 years after EUS-PCA. About 8% of patients in this trial underwent surgery for persistent cysts.

The trial will recruit patients with concerning IPMN features, for whom a multidisciplinary meeting recommends EUS-PCA as a treatment option. This patient group would usually be recommended to have surgery, but many patients decline surgery due to its high morbidity and significant mortality rates or are not candidates for this due to comorbidities or other issues. If EUS-PCA is successful, then it may ablate these precancerous lesions, treat patients who are not fit for surgery and reduce the incidence of invasive pancreatic adenocarcinoma. This is likely to reduce inequity for Māori, who are at higher risk of being ineligible for surgery for these lesions. While this is a small trial, we will also aim to recruit 50% Māori to further address inequity of opportunity and health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Radiological diagnosis of branch duct IPMN.
* Cyst size of 3cm or worrying growth on serial imaging.
* Suitable to undergo endoscopy under deep sedation or general anaesthesia.
* Willing and able to comply with all trial requirements, including treatment, timing and/or nature of required assessments.
* Signed, written informed consent.

Exclusion Criteria:

* Presence of known or suspected pancreatic cancer or pathologic lymphadenopathy.
* Radiological diagnosis of IPMN with any of the following:

  1. Main pancreatic duct dilation of >10 mm
  2. Cytology with high grade dysplasia or "suspicious for malignancy"
  3. Common bile duct obstruction causing jaundice
  4. Septated cysts with > 4 compartments
  5. Epithelial type mural nodules (> 2mm)
  6. Lesions with thick wall/septation (> 2mm)
  7. High-grade communication with the main pancreatic duct
  8. Previous aspiration failure due to excessive cyst fluid viscosity
* Clinically significant laboratory abnormalities

  1. INR >= 1.7
  2. APTT > 80 secs
  3. Platelet count < 100 x 10E9/L
  4. ALT > 500 U/L
  5. Total bilirubin > 25 umol/L
* Evidence of pancreatitis within the last 6 months.
* History of hypersensitivity to gemcitabine or paclitaxel.
* Concurrent illness that may jeopardise the ability of the patient to safely undergo the procedures outlined in this protocol.
* Any medical condition that would, at the discretion of the investigator, interfere with the completion of and/or participation in the protocol.
* Presence of any psychological, familial, sociological, or geographical condition potentially hampering compliance with the trial protocol and follow-up schedule, including alcohol dependence or drug abuse.
* Pregnancy, lactation, or inadequate contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-31 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients in whom EUS-PCA was completed as planned. | 2 years
  The proportion of patients in whom the cyst was aspirated and injected with the chemotherapy solution as intended, determined by the interventional endoscopist.

SECONDARY OUTCOMES:
The IPMN complete response rate in the injected lesion(s) on imaging 3 months post-EUS-PCA. | 2 years
  The proportion with a complete response (CR) in the injected lesion on imaging 3 months after EUS-PCA a) in all recruited patients, and b) in those in whom EUS-PCA was successfully completed.
  * The proportion with CR at 3 months in Māori and non-Māori.
  * The safety of EUS-PCA in the first 30 days post-procedure.
  * The additional resource use required for this procedure compared to EUS and cyst aspiration alone.
  * Cyst characteristics according to radiological features and amylase, CEA, viscosity, and cytology from cyst fluid.

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Jameson, PhD, Study Chair — University of Auckland, New Zealand
Locations (2):
- New Zealand (2):
  - Te Whatu Ora Waitematā, Auckland
  - Te Whatu Ora Waikato, Hamilton